CLINICAL TRIAL: NCT02716779
Title: Randomized, Multicentric, Partially Double-Blinded Placebo-Controlled Phase II Study for Examining the Influence of Ribavirin on the Initial Virological Response With Treatment of Peginterferon Alfa-2a (40KD) and Ribavirin With a Six Week Pretreatment-Phase of Ribavirin/Placebo or PEG-Interferon Monotherapy in Treatment Naïve Patients With Chronic Hepatitis C Virus Genotype 1 Infection
Brief Title: Influence of Ribavirin on the Initial Virological Response in Treatment Naïve Patients With Hepatitis C Genotype 1 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ML19301; 2006-000935-86 (EudraCT Number)
Record Dates: First submitted 2016-03-18; First posted 2016-03-23 (Estimated); Results first posted 2016-07-14 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-03

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Pegylated Interferon (PEG-IFN) alfa-2a (Experimental): Participants with chronic hepatitis C, genotype 1, received pegylated interferon (PEG-IFN) alfa-2a monotherapy for 6 weeks. Thereafter, all participants received combination therapy with PEG-IFN alfa-2a plus ribavirin for 12 weeks.
  Interventions: Drug: Pegylated Interferon (PEG-IFN) alfa-2a; Drug: Ribavirin
- Placebo (Placebo Comparator): Participants with chronic hepatitis C, genotype 1, received ribavirin matching placebo for 6 weeks. Thereafter, all participants received combination therapy with PEG-IFN alfa-2a plus ribavirin for 12 weeks.
  Interventions: Drug: Pegylated Interferon (PEG-IFN) alfa-2a; Drug: Placebo; Drug: Ribavirin
- Ribavirin (Experimental): Participants with chronic hepatitis C, genotype 1, received ribavirin monotherapy for 6 weeks. Thereafter, all participants received combination therapy with PEG-IFN alfa-2a plus ribavirin for 12 weeks.
  Interventions: Drug: Pegylated Interferon (PEG-IFN) alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Pegylated Interferon (PEG-IFN) alfa-2a — Pegylated interferon (PEG-IFN) alfa-2a (40 kilodalton [KD]) 180 microgram (mcg) subcutaneously (SC) weekly, for 6 weeks during monotherapy and/or 12 weeks during combination therapy.
  Other Names: Pegasys®
Drug: Placebo — Ribavirin matching placebo orally (PO) twice daily for 6 weeks.
  Arms: Placebo
Drug: Ribavirin — Ribavirin, 1000 mg orally (PO) (400 mg in the morning [=2 tablets] and 600 mg in the evening [=3 tablets]) in participants with a body weight less than 75 kilogram (kg) or 1200 mg PO (600 mg at each time =3 tablets, in the morning and evening, respectively) in participants with a body weight greater than or equal to 75 kg, PO daily for 6 weeks during monotherapy and/or 12 weeks during combination therapy.
  Other Names: Copegus®

SUMMARY:
This study examined the influence of ribavirin on the initial virological response in treatment-naïve participants with chronic hepatitis C, genotype 1. Participants were randomized to 1 of 3 treatment groups to receive placebo, ribavirin monotherapy 1000 milligrams (mg) to 1200 mg orally daily depending on body weight or pegylated interferon (PEG-IFN) alfa-2a (Pegasys®) 180 micrograms (mcg) subcutaneously (SC) weekly, for 6 weeks. Following the initial 6 weeks, all participants received combination therapy with PEG-IFN alfa-2a plus ribavirin (Copegus®) for 12 weeks. If there was an initial virological response after 12 weeks of combination therapy, treatment could be continued for a further 36 weeks outside of the study.

ELIGIBILITY:
Inclusion Criteria:

* Caucasians, male or female aged between 18 and 70 years
* Indication: serological proof of a chronic hepatitis C infection with positive result of anti-Hepatitis C virus (HCV) test and detectable HCV- Ribo Nucleic Acid (RNA) in serum
* Proven HCV genotype 1 by means of the reverse hybridization assays
* Proven histological infection activity within the liver with or without proven compensated cirrhosis within the last 24 months prior to start of the study (Child-Pugh degree A)
* Participants without previous anti-HCV therapy

Exclusion Criteria:

* Known hypersensitivity to interferon or ribavirin or any of the other component parts
* Pregnant or nursing women, women with child bearing potential and without using a high effective method of contraception. The urine and serum pregnancy test at visit 0 in fertile participants or cohabitants of participants must show a negative result
* Male partners of pregnant women
* Infection with HCV genotype 2, 3, 4, 5, or 6
* Pretreatment with interferon and/or ribavirin
* Immunocompromised participants
* Treatment of systemic anti-neoplastic or immunomodulatoric medication (including supraphysiological doses of steroids or radiation therapy) within the last 6 months prior to the start of treatment and during the complete time interval of study treatment
* Chronic hepatitis due to hepatitis C virus (e.g. haemochromatosis, autoimmunohepatitis, metabolic or alcohol-related liver disease)
* Decompensated liver cirrhosis or liver disease Child-Pugh degree B or C or condition after decompensation
* Signs of a hepatocellular carcinoma within 2 months prior to randomization in case of a cirrhosis or a transition to cirrhosis
* Ascites or esophagus varices with bleedings as documented in anamnesis
* Any medical condition that questions in the opinion of the investigator the participant's enrollment and participation in the trial
* Hemoglobin <13 grams/deciliter (g/dl) in females and <14 g/dl in males in screening phase
* Patients with an increased anemia risk (e.g. thalassemia, spherocytosis, etc.) or patients which would be at a particular medical risk in case of an anemia
* Diagnosed neutropenia <1.500/microliter (mcl) or thrombocytopenia <90.000/mcl in screening phase

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Zeuzem, Prof. Dr., Principal Investigator — Roche Pharma AG, 79639 Grenazch Wyhlen, Germany
Locations (4):
- Germany (4):
  - Berlin
  - Frankfurt am Main
  - Hanover
  - Homburg/ Saar

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment was 68: 1 participant withdrew during the screening phase and 67 participants were randomized.
Groups:
- Placebo: Participants with chronic hepatitis C, genotype 1, received ribavirin matching placebo for 6 weeks. Thereafter, all participants received combination therapy with PEG-IFN alfa-2a plus ribavirin for 12 weeks.
  Pegylated Interferon (PEG-IFN) alfa-2a: Pegylated Interferon (PEG-IFN) alfa-2a (40 kilodalton [KD]) 180 microgram (mcg) subcutaneously (SC) weekly, for 6 weeks during monotherapy and/or 12 weeks during combination therapy.
  Placebo: Ribavirin matching placebo orally (PO) twice daily for 6 weeks.
  Ribavirin: Ribavirin, 1000 mg PO (400 mg in the morning [=2 tablets] and 600 mg in the evening [=3 tablets]) in participants with a body weight less than 75 kilogram (kg) or 1200 mg PO (600 mg at each time =3 tablets, in the morning and evening, respectively) in participants with a body weight greater than or equal to 75 kg, PO daily for 6 weeks during monotherapy and/or 12 weeks during combination therapy.
Period: Monotherapy
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a | Placebo | Ribavirin
Started | 14 | 26 | 27
Completed | 14 | 25 | 26
Not Completed | 0 | 1 | 1
Not completed — Adverse Event | 0 | 1 | 1
Period: Combination Therapy
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a | Placebo | Ribavirin
Started | 14 | 25 | 26
Completed | 14 | 23 | 25
Not Completed | 0 | 2 | 1
Not completed — Adverse Event | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Pegylated Interferon (PEG-IFN) Alfa-2a: Participants with chronic hepatitis C, genotype 1, received pegylated interferon (PEG-IFN) alfa-2a monotherapy for 6 weeks. Thereafter, all participants received combination therapy with PEG-IFN alfa-2a plus ribavirin for 12 weeks.
  Pegylated Interferon (PEG-IFN) alfa-2a: Pegylated Interferon (PEG-IFN) alfa-2a (40KD) 180 microgram (mcg) subcutaneously (SC) weekly, for 6 weeks during monotherapy and/or 12 weeks during combination therapy.
  Ribavirin: Ribavirin, 1000 mg PO (400 mg in the morning [=2 tablets] and 600 mg in the evening [=3 tablets]) in participants with a body weight less than 75 kilogram (kg) or 1200 mg PO (600 mg at each time =3 tablets, in the morning and evening, respectively) in participants with a body weight greater than or equal to 75 kg, PO daily for 6 weeks during monotherapy and/or 12 weeks during combination therapy.
- Placebo: Participants with chronic hepatitis C, genotype 1, received ribavirin matching placebo for 6 weeks. Thereafter, all participants received combination therapy with PEG-IFN alfa-2a plus ribavirin for 12 weeks.
  Pegylated Interferon (PEG-IFN) alfa-2a: Pegylated Interferon (PEG-IFN) alfa-2a (40KD) 180 microgram (mcg) subcutaneously (SC) weekly, for 6 weeks during monotherapy and/or 12 weeks during combination therapy.
  Placebo: Ribavirin matching placebo orally (PO) twice daily for 6 weeks.
  Ribavirin: Ribavirin, 1000 mg PO (400 mg in the morning [=2 tablets] and 600 mg in the evening [=3 tablets]) in participants with a body weight less than 75 kilogram (kg) or 1200 mg PO (600 mg at each time =3 tablets, in the morning and evening, respectively) in participants with a body weight greater than or equal to 75 kg, PO daily for 6 weeks during monotherapy and/or 12 weeks during combination therapy.
- Ribavirin: Participants with chronic hepatitis C, genotype 1, received ribavirin monotherapy for 6 weeks. Thereafter, all participants received combination therapy with PEG-IFN alfa-2a plus ribavirin for 12 weeks.
  Pegylated Interferon (PEG-IFN) alfa-2a: Pegylated Interferon (PEG-IFN) alfa-2a (40KD) 180 microgram (mcg) subcutaneously (SC) weekly, for 6 weeks during monotherapy and/or 12 weeks during combination therapy.
  Ribavirin: Ribavirin, 1000 mg PO (400 mg in the morning [=2 tablets] and 600 mg in the evening [=3 tablets]) in participants with a body weight less than 75 kilogram (kg) or 1200 mg PO (600 mg at each time =3 tablets, in the morning and evening, respectively) in participants with a body weight greater than or equal to 75 kg, PO daily for 6 weeks during monotherapy and/or 12 weeks during combination therapy.
- Total: Total of all reporting groups
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a | Placebo | Ribavirin | Total
Number analyzed (Participants) | 14 | 26 | 27 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (14.4) | 48.2 (15.4) | 50.2 (12.9) | 48.5 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 18 | 17 | 42
  Male | 7 | 8 | 10 | 25

OUTCOME MEASURES:

1. Primary Outcome: Log Likelihood Median Values of Hepatitis C-Virus (HCV) Kinetic Models for Quantitative HCV Ribonucleic Acid (RNA) Measurement With Various Assumptions of Ribavirin Mechanism of Action
Description: To investigate possible action mechanisms, three different models were fitted to viruskinetic data and evaluated using related log-likelihood function values. These models were designed assuming individual effects with respect to infectiousness (model 1), virus production (model 2) or degradation of infected cells rate (model 3). The following viruskinetic parameters were fitted in each model: initial viral load, loss rate of infected cells (delta), effectivity of interferon with respect to a pharmacokinetic-pharmacodynamic model. A lower log likelihood function value indicates a lesser fit for the model.
Time Frame: Up to Day 126
Population: Per Protocol (PP) population: participants with 6 weeks of monotherapy and at least 4 weeks combination therapy as well as three quantitative HCV-RNA measurements (baseline, period 1, period 2), no major protocol violations, no treatment interruption and no dose reduction below 80% of the planned medication within the first 10 therapy weeks.
Measure: Median (95% Confidence Interval); unit: log likelihood function value
Groups:
- Total Participant Group: Combined group of PEG IFN alfa-2a, matching placebo and ribavirin arms.
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a | Ribavirin | Total Participant Group
Number analyzed (Participants) | 13 | 23 | 61
log likelihood function value
  Model 1= infectiousness | -27.0 [-34.5 to -14.0] | -21.4 [-24.7 to -15.2] | -22.2 [-26.0 to -19.3]
  Model 2= virus production | -28.2 [-35.0 to -14.3] | -23.8 [-27.5 to -21.6] | -23.9 [-27.4 to -21.6]
  Model 3= degradation rate | -27.1 [-33.2 to -14.0] | -20.7 [-25.5 to -16.0] | -23.1 [-26.5 to -18.4]

2. Secondary Outcome: Score in Quality of Life Assessed Using Short Form-36 (SF-36) Health Questionnaire
Description: SF-36 is a psychometric scale to quantify health conditions. This psychometric scale has 8 dimensions of the subjective health status and consists of 36 individual items that have a varying number of related item scores (ranging from "yes/no" up to a 6-point scale). At first the raw scores were determined by summation over all items and weighted accordingly. Afterwards the raw scores were transformed to ranges of 0-100 with 100 being the highest level of health and compared to published reference scales. The following eight dimensions of subjective health conditions were considered: physical functioning index, role physical index, pain, general health perception, vitality, social functioning index, role emotional index and mental health index. The SF36 questionnaire had to be answered by the patients at screening before monotherapy, after monotherapy and at the end of the study (=end of combination therapy).
Time Frame: At screening (Days -56 to -1), at end of monotherapy (Week 6) and at end of combination therapy (Week 18)
Population: Intent-to-treat (ITT) population includes all randomized participants who received at least one dose of study drug. Here, 'n' is the number of evaluable participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a | Placebo | Ribavirin
Number analyzed (Participants) | 6 | 11 | 17
units on a scale
  Physical functioning index: Screening | 95.6 (5.2) | 76.5 (20.2) | 79.7 (28.7)
  Physical functioning index: End of monotherapy | 90.8 (9.2) | 72.3 (28.1) | 68.4 (27.7)
  Physical functioning index: End of comb. therapy | 67.1 (20.7) | 73.0 (14.0) | 53.4 (31.5)
  Role physical index: Screening | 75.0 (41.8) | 55.6 (41.0) | 62.5 (40.8)
  Role physical index: End of monotherapy | 66.7 (34.2) | 56.8 (43.4) | 50.5 (40.5)
  Role physical index: End of combination therapy | 25.0 (38.7) | 40.0 (35.7) | 29.7 (40.0)
  Pain: Screening | 89.3 (17.0) | 70.3 (26.8) | 70.0 (30.8)
  Pain: End of monotherapy | 73.2 (23.3) | 61.5 (27.4) | 66.0 (29.6)
  Pain: End of combination therapy | 72.3 (32.2) | 56.0 (11.8) | 60.1 (34.8)
  General health perception: Screening | 58.6 (12.9) | 53.6 (14.5) | 62.9 (14.5)
  General health perception: End of monotherapy | 58.2 (7.6) | 59.2 (16.9) | 54.3 (18.0)
  General health perception: End of comb. therapy | 60.0 (14.3) | 55.2 (15.0) | 47.1 (20.6)
  Vitality: Screening | 54.2 (9.2) | 52.8 (21.5) | 50.9 (18.9)
  Vitality: End of monotherapy | 45.0 (15.2) | 44.1 (16.3) | 41.8 (20.1)
  Vitality: End of combination therapy | 40.8 (14.6) | 32.5 (12.1) | 39.8 (16.1)
  Social functioning index: Screening | 75.0 (23.7) | 79.2 (24.2) | 83.8 (20.6)
  Social functioning index: End of monotherapy | 72.9 (22.9) | 68.2 (24.0) | 80.1 (22.6)
  Social functioning index: End of comb. therapy | 68.8 (23.4) | 61.3 (19.9) | 56.3 (25.8)
  Role emotional index: Screening | 55.6 (50.2) | 66.7 (50.0) | 62.5 (43.7)
  Role emotional index: End of monotherapy | 55.6 (50.2) | 69.7 (45.8) | 53.3 (51.6)
  Role emotional index: End of combination therapy | 33.3 (51.6) | 50.0 (42.3) | 35.4 (39.4)
  Mental health index: Screening | 68.5 (9.1) | 63.1 (18.1) | 64.5 (15.4)
  Mental health index: End of monotherapy | 61.3 (12.3) | 62.8 (14.0) | 61.5 (19.7)
  Mental health index: End of combination therapy | 72.2 (9.0) | 61.6 (13.2) | 47.7 (23.0)

3. Secondary Outcome: Percentage of Participants With Treatment Response
Description: HCV-RNA level was measured at each visit by a central laboratory. Treatment response was estimated applying the following definitions of response/non-response: 1) Adequate first phase decline: HCV RNA decline ≥ 0.5 log10 International Units/milliliter (IU/mL) from time 0 to 48 hours of PEG-IFN treatment (PEG-IFN arm: day 0 - day 2; placebo and ribavirin arm: day 42-day 44), 2) Rapid virologic response: HCV RNA < 15 IU/mL (=detection limit) on day 70, 3) Complete early virologic response: HCV RNA < 15 IU/mL on day 126, 4) Partial early virologic response (log decrease): HCV RNA decrease ≥ 2 log10 IU/mL from day 0 to day 126, 5) Partial early virologic response (cut off): HCV RNA <30000 IU/mL on day 126, 6) Non-response: HCV RNA decrease <2 log10 IU/mL from day 0 to day 126, 7) Null-response: HCV RNA decrease <1 log10 IU/mL from day 0 to day 28 and from day 0 to day 70 for PEG-IFN arm and placebo / ribavirin arm, respectively.
Time Frame: Up to Day 126
Population: All evaluable participants of the Intent-to-Treat (ITT) population, who were documented for a total of 126 days of the treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a | Placebo | Ribavirin
Number analyzed (Participants) | 14 | 23 | 25
percentage of participants
  Adequate first phase decline | 79 | 65 | 72
  Rapid virologic response | 43 | 30 | 20
  Complete early virologic response | 64 | 48 | 72
  Partial early virologic response (log decrease) | 79 | 78 | 84
  Partial early virologic response (cut off) | 79 | 78 | 84
  Non-response | 21 | 22 | 16
  Null responder | 36 | 26 | 12

4. Secondary Outcome: Area Under the Concentration-Time Curve (AUC) of Ribavirin
Description: Evaluation of ribavirin arm after Day 0. Evaluation of placebo and PEG-IFN arms after Day 42.
Time Frame: From Day 0 at 0 hour (hr), 12 hr, 24 hr, 36 hr, 48 hr, 60 hr and 72 hr, Day 42 at 0 hr, 12 hr, 24 hr and 36 hr and at each visit up to Day 126.
Population: All evaluable participants of the ITT population, who were documented for a total of 126 days of the treatment period.
Measure: Median (95% Confidence Interval); unit: (microgram/milliliter)*day ([mcg/ml]*d)
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a | Placebo | Ribavirin
Number analyzed (Participants) | 13 | 23 | 25
(microgram/milliliter)*day ([mcg/ml]*d) | 186.6 [142.3 to 201.4] | 179.4 [142.6 to 203.8] | 290.1 [257.6 to 370.5]

5. Secondary Outcome: Maximum Concentration (Cmax) of Ribavirin
Description: Cmax was obtained directly from the concentration-time data. Evaluation of ribavirin arm after day 0. Evaluation of placebo and PEG-IFN arms after day 42.
Time Frame: as for outcome 4
Population: All evaluable participants of the ITT population, who were documented for a total of 126 days of the treatment period.
Measure: Median (95% Confidence Interval); unit: mcg/ml
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a | Placebo | Ribavirin
Number analyzed (Participants) | 13 | 23 | 25
mcg/ml | 2.95 [2.79 to 3.60] | 2.83 [2.34 to 3.26] | 3.37 [2.93 to 4.19]

6. Secondary Outcome: Time to Maximum Concentration (Tmax) of Ribavirin
Description: Tmax was obtained directly from the concentration-time data. Evaluation of ribavirin arm after day 0. Evaluation of placebo and PEG-IFN arms after day 42.
Time Frame: as for outcome 4
Population: All evaluable participants of the ITT population, who were documented for a total of 126 days of the treatment period.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a | Placebo | Ribavirin
Number analyzed (Participants) | 13 | 23 | 25
weeks | 6.0 [4.0 to 12.0] | 8.0 [6.0 to 12.0] | 6.4 [6.1 to 8.0]

7. Secondary Outcome: Area Under the Concentration-Time Curve (AUC) of PEG-IFN
Description: Evaluation of PEG-IFN arm after Day 0. Evaluation of ribavirin and placebo arms after Day 42.
Time Frame: From Day 0 at 0 hour (hr), 24 hr, 48 hr and 72 hr, Day 42 at 0 hr and 24 hr and at approximately every other visit up to Day 126
Population: All evaluable participants of the ITT population, who were documented for a total of 126 days of the treatment period.
Measure: Median (95% Confidence Interval); unit: (nanogram/milliliter)*day ([ng/ml]*d)
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a | Placebo | Ribavirin
Number analyzed (Participants) | 14 | 22 | 25
(nanogram/milliliter)*day ([ng/ml]*d) | 2097.9 [1763.5 to 2997.3] | 1270.4 [931.8 to 1572.0] | 1164.9 [925.2 to 1461.3]

8. Secondary Outcome: Maximum Concentration (Cmax) of PEG-IFN
Description: Cmax was obtained directly from the concentration-time data. Evaluation of PEG-IFN arm after day 0. Evaluation of ribavirin and placebo arms after day 42.
Time Frame: as for outcome 7
Population: All evaluable participants of the ITT population, who were documented for a total of 126 days of the treatment period.
Measure: Median (95% Confidence Interval); unit: ng/ml
Groups:
- Placebo: Participants with chronic hepatitis C, genotype 1, received ribavirin matching placebo monotherapy for 6 weeks. Thereafter, all participants received combination therapy with PEG-IFN alfa-2a plus ribavirin for 12 weeks.
  Pegylated Interferon (PEG-IFN) alfa-2a: Pegylated Interferon (PEG-IFN) alfa-2a (40KD) 180 microgram (mcg) subcutaneously (SC) weekly, for 6 weeks during monotherapy and/or 12 weeks during combination therapy.
  Placebo: Ribavirin matching placebo orally (PO) twice daily for 6 weeks.
  Ribavirin: Ribavirin, 1000 mg PO (400 mg in the morning [=2 tablets] and 600 mg in the evening [=3 tablets]) in participants with a body weight less than 75 kilogram (kg) or 1200 mg PO (600 mg at each time =3 tablets, in the morning and evening, respectively) in participants with a body weight greater than or equal to 75 kg, PO daily for 6 weeks during monotherapy and/or 12 weeks during combination therapy.
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a | Placebo | Ribavirin
Number analyzed (Participants) | 14 | 22 | 25
ng/ml | 28.77 [22.80 to 32.38] | 20.36 [16.92 to 25.83] | 19.8 [15.80 to 22.30]

9. Secondary Outcome: Time to Maximum Concentration (Tmax) of PEG-IFN
Description: Tmax was obtained directly from the concentration-time data. Evaluation of PEG-IFN arm after day 0. Evaluation of ribavirin and placebo arms after day 42.
Time Frame: as for outcome 7
Population: All evaluable participants of the ITT population, who were documented for a total of 126 days of the treatment period.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a | Placebo | Ribavirin
Number analyzed (Participants) | 14 | 22 | 25
weeks | 6.3 [6.1 to 8.0] | 12.0 [6.0 to 12.0] | 6.0 [6.0 to 12.0]

10. Secondary Outcome: Area Under the Concentration-Time Curve (AUC) of Glutamate-Pyruvate Transaminase (GPT)
Time Frame: as for outcome 4
Population: All evaluable participants of the ITT population, who were documented for a total of 126 days of the treatment period.
Measure: Median (95% Confidence Interval); unit: (Units/liter)*day ([U/L]*d)
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a | Placebo | Ribavirin
Number analyzed (Participants) | 14 | 23 | 25
(Units/liter)*day ([U/L]*d) | 5078.3 [4358.3 to 6576.5] | 7233.5 [5337.3 to 8656.3] | 5231.3 [3917.0 to 5852.5]

11. Secondary Outcome: Maximum Concentration (Cmax) of GPT
Description: Cmax was obtained directly from the concentration-time data.
Time Frame: as for outcome 4
Population: All evaluable participants of the ITT population, who were documented for a total of 126 days of the treatment period.
Measure: Median (95% Confidence Interval); unit: U/L
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a | Placebo | Ribavirin
Number analyzed (Participants) | 14 | 23 | 25
U/L | 68.5 [59.0 to 112.0] | 88.0 [67.0 to 123.0] | 75.0 [56.0 to 110.0]

12. Secondary Outcome: Time to Maximum Concentration (Tmax) of GPT
Description: Tmax was obtained directly from the concentration-time data.
Time Frame: as for outcome 4
Population: All evaluable participants of the ITT population, who were documented for a total of 126 days of the treatment period.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pegylated Interferon (PEG-IFN) Alfa-2a | Placebo | Ribavirin
Number analyzed (Participants) | 14 | 23 | 25
days | 2.8 [2.0 to 28.0] | 14.0 [10.0 to 42.5] | 3.0 [2.0 to 7.0]

ADVERSE EVENTS:
Time Frame: Up to Day 126
Groups:
- PEG-IFN Alfa-2a, Period 1 Monotherapy: Participants with chronic hepatitis C, genotype 1, received pegylated interferon (PEG-IFN) alfa-2a monotherapy for 6 weeks in period 1.
  Pegylated Interferon (PEG-IFN) alfa-2a: Pegylated Interferon (PEG-IFN) alfa-2a (40KD) 180 microgram (mcg) subcutaneously (SC) weekly, for 6 weeks.
- Placebo, Period 1 Monotherapy: Participants with chronic hepatitis C, genotype 1, received placebo PO for 6 weeks in period 1.
  Placebo: Ribavirin matching placebo orally (PO) twice daily for 6 weeks.
- Ribavirin, Period 1 Monotherapy: Participants with chronic hepatitis C, genotype 1, received ribavirin monotherapy for 6 weeks in period 1.
  Ribavirin: Ribavirin, 1000 mg PO (400 mg in the morning [=2 tablets] and 600 mg in the evening [=3 tablets]) in participants with a body weight less than 75 kilogram (kg) or 1200 mg PO (600 mg at each time =3 tablets, in the morning and evening, respectively) in participants with a body weight greater than or equal to 75 kg, PO daily for 6 weeks.
- PEG-IFN Alfa-2a, Period 2 Combination Therapy: In period 2 participants, who received PEG-IFN monotherapy in period 1, received combination therapy with PEG-IFN alfa-2a plus ribavirin for 12 weeks.
  Pegylated Interferon (PEG-IFN) alfa-2a: Pegylated Interferon (PEG-IFN) alfa-2a (40KD) 180 microgram (mcg) subcutaneously (SC) weekly, for 6 weeks.
  Ribavirin: Ribavirin, 1000 mg PO (400 mg in the morning [=2 tablets] and 600 mg in the evening [=3 tablets]) in participants with a body weight less than 75 kilogram (kg) or 1200 mg PO (600 mg at each time =3 tablets, in the morning and evening, respectively) in participants with a body weight greater than or equal to 75 kg, PO daily for 6 weeks.
- Placebo, Period 2 Combination Therapy: In period 2 participants, who received placebo in period 1, received combination therapy with PEG-IFN alfa-2a plus ribavirin for 12 weeks.
  Pegylated Interferon (PEG-IFN) alfa-2a: Pegylated Interferon (PEG-IFN) alfa-2a (40KD) 180 microgram (mcg) subcutaneously (SC) weekly, for 6 weeks.
  Ribavirin: Ribavirin, 1000 mg PO (400 mg in the morning [=2 tablets] and 600 mg in the evening [=3 tablets]) in participants with a body weight less than 75 kilogram (kg) or 1200 mg PO (600 mg at each time =3 tablets, in the morning and evening, respectively) in participants with a body weight greater than or equal to 75 kg, PO daily for 6 weeks.
- Ribavirin, Period 2 Combination Therapy: In period 2 participants, who received ribavirin monotherapy in period 1, received combination therapy with PEG-IFN alfa-2a plus ribavirin for 12 weeks.
  Pegylated Interferon (PEG-IFN) alfa-2a: Pegylated Interferon (PEG-IFN) alfa-2a (40KD) 180 microgram (mcg) subcutaneously (SC) weekly, for 6 weeks.
  Ribavirin: Ribavirin, 1000 mg PO (400 mg in the morning [=2 tablets] and 600 mg in the evening [=3 tablets]) in participants with a body weight less than 75 kilogram (kg) or 1200 mg PO (600 mg at each time =3 tablets, in the morning and evening, respectively) in participants with a body weight greater than or equal to 75 kg, PO daily for 6 weeks.
Arm/Group | PEG-IFN Alfa-2a, Period 1 Monotherapy | Placebo, Period 1 Monotherapy | Ribavirin, Period 1 Monotherapy | PEG-IFN Alfa-2a, Period 2 Combination Therapy | Placebo, Period 2 Combination Therapy | Ribavirin, Period 2 Combination Therapy
Serious Adverse Events (participants affected / at risk) | 0/14 | 1/26 | 0/27 | 0/14 | 2/25 | 2/26
Other Adverse Events (participants affected / at risk) | 9/14 | 9/26 | 12/27 | 12/14 | 23/25 | 24/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-IFN Alfa-2a, Period 1 Monotherapy (N=14) | Placebo, Period 1 Monotherapy (N=26) | Ribavirin, Period 1 Monotherapy (N=27) | PEG-IFN Alfa-2a, Period 2 Combination Therapy (N=14) | Placebo, Period 2 Combination Therapy (N=25) | Ribavirin, Period 2 Combination Therapy (N=26)
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Psychotherapy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-IFN Alfa-2a, Period 1 Monotherapy (N=14) | Placebo, Period 1 Monotherapy (N=26) | Ribavirin, Period 1 Monotherapy (N=27) | PEG-IFN Alfa-2a, Period 2 Combination Therapy (N=14) | Placebo, Period 2 Combination Therapy (N=25) | Ribavirin, Period 2 Combination Therapy (N=26)
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Keratoconjunctivitis sicca (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 1 | 4 | 8 | 5
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 5 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Fatigue (General disorders) | 3 | 1 | 4 | 0 | 9 | 6
Chills (General disorders) | 2 | 1 | 0 | 0 | 3 | 1
Influenza like illness (General disorders) | 3 | 0 | 0 | 1 | 5 | 9
Asthenia (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 1 | 3 | 3
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 4 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 2 | 2 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1
Headache (Nervous system disorders) | 2 | 4 | 4 | 2 | 10 | 5
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 5
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 2
Sleep disorder (Psychiatric disorders) | 0 | 1 | 2 | 0 | 4 | 2
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0
Initial insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 2 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 5 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 2 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.